CLINICAL TRIAL: NCT05065736
Title: 18F-Clofarabine (CFA) as a PET Imaging Agent to Measure Deoxycytidine Kinase (DCK) Activity in Metastatic Cancer, as a Candidate Predictive Biomarker for Response to DCK-dependent Drugs Such as Gemcitabine
Brief Title: Using a PET Imaging Agent, 18F-Clofarabine (CFA), to Measure Deoxycytidine Kinase Activity in Metastatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roberto Vargas (Other)
Responsible Party: Sponsor-Investigator, Roberto Vargas, PI, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE4Y21
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Cancer; Carcinoma; Adenocarcinoma
Keywords: 18F-Clofarabine; Diagnostic Imaging; Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma; Adenocarcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-Clofarabine (Experimental): 18F-Clofarabine as PET imaging agent for measuring the activity of deoxycytidine kinase (DCK) in various normal and abnormal tissues in cancer participants before and after therapy
  Interventions: Drug: 18F-Clofarabine

INTERVENTIONS:
Drug: 18F-Clofarabine — The participants enrolled will receive a baseline CFA PET/CT evaluation. Then, the participants will undergo the routine follow up would normally occur for their cancer and its treatment. If this routine follow up and care involves repeat imaging of the cancer, then the CFA PET/CT scan will be repeated at that time (timed according to standard-of-care follow-up imaging), which is expected between a month to about 4 months after the first CFA PET/CT scan. The study period will end 24 hours after this repeat PET/CT scan.

SUMMARY:
The purpose of this study is to evaluate whether a new type of imaging study, called 18F-Clofarabine (CFA) PET/CT, can be used to image cancer pyrimidine metabolism in participants.

PET (positron emission tomography) imaging is a way of looking at cancers that can reveal cancer metabolism. Presently, however, there are no imaging agents in routine use to look at an aspect of cancer metabolism (pyrimidine metabolism) that dictates whether certain cancer drugs, e.g., gemcitabine, are likely to be taken into the cancer cells. This clinical trial will be testing whether 18F-Clofarabine (CFA) could be an imaging agent to measure this aspect of cancer metabolism.

DETAILED DESCRIPTION:
The participants will receive a CFA injection into a vein in their arm. The imaging drug is attracted to and taken into certain cells in the body, including cancer cells. 18F-Clofarabine (CFA) is experimental because it is not approved by the Food and Drug Administration (FDA).

The participants will be observed for side effects, and about 1 hour later, they will receive a PET/CT scan. Additionally, they will be contacted the next day to inquire again about any side effects. If the participant's routine care involves repeat imaging of cancer, then the CFA PET/CT scan will be repeated at that time, which could be up to 365 days after the first CFA PET/CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven metastatic cancer (including carcinoma, adenocarcinoma, sarcoma, or neuroendocrine cancer).
* Subjects must have metastatic disease, confirmed by imaging, typically a CT scan of the chest/abdomen/pelvis.
* Subjects must have measurable disease per RECIST 1.1
* Over 18 years of age
* ECOG performance status 0-1
* Adequate organ function as defined by the following criteria (labs may be no more than 4 weeks prior to the screening date):

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) <= 2.5 x laboratory upper limit of normal (ULN)
  * Total serum bilirubin <= 2.0 x ULN
  * Absolute neutrophil count (ANC) >= 1500/uL
  * Platelets >= 75,000/uL
  * Hemoglobin >= 8.0 g/dL
  * Serum calcium <= 12.0 mg/dL
  * Serum creatinine <= 2.9 mg/dL
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Patient is able to remain still for the duration of the imaging procedure (up to one hour).

Exclusion Criteria:

* Within 6 months prior to enrollment on this study: myocardial infarction, severe/unstable angina, severe peripheral vascular disease (claudication) or procedure on peripheral vasculature, coronary/peripheral artery bypass graft, New York Heart Association grade II or greater congestive heart failure, cerebrovascular accident or transient ischemic attack, clinically significant bleeding or pulmonary embolism.
* Pregnancy or breastfeeding (pregnant or breastfeeding women are excluded from this study because study drugs have the potential for teratogenic or abortifacient effects.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate CFA as a PET imaging agent | up to 60 minutes after CFA PET
  Establish the image-based biodistribution of CFA, a new tracer for imaging DCK enzyme activity. DCK converts the inactive prodrug clofarabine into its active form. Thus, the degree of DCK expression in normal and abnormal tissues may predict drug effects and effectiveness.
  The uptake of the radiotracer (SUVs) will be measured quantitatively from PET images taken at 60 min post-injection of [18F]CFA.

SECONDARY OUTCOMES:
Correlate CFA uptake with conventional imaging | up to 3 months after CFA PET
  Correlate CFA uptake with conventional anatomic imaging using RECIST criteria to establish change over time and differences from participants' baseline scans.
Correlate CFA uptake with PFS | up to 12 months after CFA PET
  Correlate changes in CFA uptake (SUV) with disease progression as determined by standard of care surveillance imaging.
Correlate CFA uptake with OS | up to 12 months after CFA PET
  Correlate changes in CFA uptake with participant outcomes as measured by all cause mortality/overall survival (OS).
Adverse Events | within 48 hrs of radiotracer administration
  Proportion of participants who develop any side effects/adverse events associated with radiotracer infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Vargas, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study of a novel PET-scan imaging agent and IPD is not needed for interpretation of the data